CLINICAL TRIAL: NCT02097771
Title: Gastric Insufflation and Laryngeal Mask Airway
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lionel Bouvet (Other)
Responsible Party: Sponsor-Investigator, Lionel Bouvet, MD PhD, Hôpital Edouard Herriot
Organization: Hôpital Edouard Herriot (Other)
Allocation: Randomized
Other Study IDs: 2013-A01852-43
Record Dates: First submitted 2014-03-21; First posted 2014-03-27 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Gastric Insufflation
Keywords: laryngeal mask airway ventilation

ARMS (2):
- LMA SupremeTM (Active Comparator)
  Interventions: Device: LMA SupremeTM
- Ambu AuraOnce (Sham Comparator)
  Interventions: Device: AuraOnceTM

INTERVENTIONS:
Device: LMA SupremeTM
  Arms: LMA SupremeTM
Device: AuraOnceTM
  Arms: Ambu AuraOnce

SUMMARY:
Comparison of the incidence of gastric insufflation between two kinds of laryngeal masks airways: LMA SupremeTM vs Ambu AuraOnceTM

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 or 2
* Age > 18 yrs
* Use of laryngeal mask airway required

Exclusion Criteria:

* risk of pulmonary aspiration of gastric contents
* Contraindication for the use of laryngeal mask airway
* Tracheal intubation required
* Patient's refusal

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2014-11; Primary Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
incidence of gastric insufflation | during pulmonary ventilation through the laryngeal mask airway

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon, France